CLINICAL TRIAL: NCT04837404
Title: Ultrasound Guided Transfemoral Complex Large-bore PCI Trial
Acronym: ULTRACOLOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maatschap Cardiologie Zwolle (Other)
Collaborators: Diagram B.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9343
Record Dates: First submitted 2021-03-01; First posted 2021-04-08 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Complex Coronary Lesions; Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre, randomized investigator-initiated trial with a superiority design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided femoral access (Other): Patients who are planned for complex PCI requiring 7 or more French sheath and guiding catheters. Ultrasound guided femoral access will be used.
  Interventions: Procedure: Ultrasound guided femoral access for complex PCI
- fluoroscopy guided femoral access (Other): Patients who are planned for complex PCI requiring 7 or more French sheath and guiding catheters. Fluoroscopy guided femoral access will be used.
  Interventions: Procedure: Fluoroscopy guided femoral access for complex PCI

INTERVENTIONS:
Procedure: Ultrasound guided femoral access for complex PCI — Ultrasound guided femoral access for complex PCI
  Arms: ultrasound guided femoral access
Procedure: Fluoroscopy guided femoral access for complex PCI — Fluoroscopy guided femoral access for complex PCI
  Arms: fluoroscopy guided femoral access

SUMMARY:
ULTRACOLOR is a randomized multicentre investigator-initiated study to investigate if ultrasound guided femoral access is associated with less clinically relevant access site related bleeding and/or vascular complications requiring intervention as compared to the fluoroscopy guided method for complex PCI with large-bore access.

DETAILED DESCRIPTION:
ULTRACOLOR is a prospective, multicentre, randomized investigator-initiated trial designed to enroll 542 subjects with an indication for PCI for complex coronary lesions.

This study will investigate if ultrasound guided femoral access is associated with less clinically relevant access site related bleeding and/or vascular complications requiring intervention as compared to the fluoroscopy guided method for complex PCI with large-bore access.

ELIGIBILITY:
Inclusion Criteria:

1. Use of the femoral artery for primary or secondary access with ≥ 7 Fr guiding catheter as indication for complex PCI, according to the expertise of the treating physician.
2. Age 18 years or older.

Exclusion Criteria:

1. Inability to obtain informed consent
2. Contra-indication for femoral access
3. Cardiogenic shock
4. ST elevation myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with BARC 2, 3 or 5 access-site related bleeding or vascular complication requiring intervention of the primary femoral access site during index hospitalization. | up to discharge hospital, on average 24 hours

SECONDARY OUTCOMES:
Proportion of patients with BARC 2, 3 or 5 access-site related bleeding or vascular complication requiring intervention of the secondary femoral or radial access site during index hospitalization. | up to discharge hospital, on average 24 hours
Proportion of patients with BARC 2, 3 or 5 access-site related bleeding or vascular complication requiring intervention of the primary femoral access site at 1 month. | 1 month
Proportion of patients with BARC 2, 3 or 5 access-site related bleeding or vascular complication requiring intervention of the secondary femoral or radial access site at 1 month | 1 month
Proportion of patients with MACE | up to discharge hospital (on average 24 hours) and at 1 month
Procedural duration | during PCI procedure
Incidence of first pass puncture | during PCI procedure
Number of access attempts | during PCI procedure
Incidence of.accidental venipuncture | during PCI procedure
Incidence of access below the femoral artery bifurcation (ileofemoral angiogram) | during PCI procedure
Incidence of vascular complication not requiring intervention of the primary femoral access site | up to discharge hospital (on average 24 hours) and at 1 month
Incidence of vascular complication not requiring intervention of the secondary femoral or radial access site | up to discharge hospital (on average 24 hours) and at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van Leeuwen, MD, PhD, Principal Investigator — Isala
Locations (10):
- Belgium (3):
  - CHU Charleroi, Charleroi
  - Ziekenhuis Oost Limburg, Genk
  - Jessa hospital, Hasselt
- Elisabeth-Krankenhaus, Essen, Germany
- Netherlands (6):
  - Amsterdam UMC, Amsterdam
  - Catharina hospital, Eindhoven
  - St Antonius, Nieuwegein
  - Radboudumc, Nijmegen
  - UMC Utrecht, Utrecht
  - Isala Hospital, Zwolle

REFERENCES:
- [Derived] Meijers TA, Nap A, Aminian A, Schmitz T, Dens J, Teeuwen K, van Kuijk JP, van Wely M, Bataille Y, Kraaijeveld AO, Roolvink V, Dambrink JE, Gosselink ATM, Hermanides RS, Ottervanger JP, Tsilingiris I, van den Buijs DMF, van Royen N, van Leeuwen MAH. Ultrasound-guided versus fluoroscopy-guided large-bore femoral access in PCI of complex coronary lesions: the international, multicentre, randomised ULTRACOLOR Trial. EuroIntervention. 2024 Jul 15;20(14):e876-e886. doi: 10.4244/EIJ-D-24-00089. PMID 38742577